CLINICAL TRIAL: NCT00212641
Title: Randomized Double-Blind Placebo-Controlled Pharmacodynamic Evaluation of ONO-5129 in Patients With Treatment Naive Type 2 Diabetes Mellitus
Brief Title: A Phase II Study to Evaluate the Effects of Oral ONO-5129 in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5129POU006
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: ONO-5129

SUMMARY:
The objectives of this study are to characterize the pharmacodynamic profile, safety and tolerability of ONO-5129 in patients with Type 2 Diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 Diabetes Mellitus
2. FBG level > 140 mg/dL and < 270 mg/dL
3. Fasting TG level < 500 mg/dL
4. BMI of 22 to 40 kg/m2, inclusive
5. Other Inclusion criteria as specified in the study protocol

Exclusion Criteria:

1. Previous participation in an ONO-5129 protocol
2. Previous treatment with TZD agents or other current antidiabetics
3. History of myocardial infarction, coronary artery surgery, atrial/ventricular tachycardia, or atrial/ventricular fibrillation in the past six months
4. Presence of functional limitations due to cardiovascular disease in accordance with the New York Heart Association Classification System - Class III (moderate) or IV (severe)
5. Other exclusion criteria as specified in the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105
Dates: Start 2005-06; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose at 8 weeks

SECONDARY OUTCOMES:
Pharmacodynamic parameters at all time points

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G Bisaha, Ph.D., Study Director — Ono Pharma USA Inc
Locations (67):
- United States (67):
  - Apex Clinical Trials, Inc., Birmingham, Alabama
  - Greystone Medical Research, LLC, Birmingham, Alabama
  - Med Search, LLC, Calera, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Clinic of Physicians and Surgeons, Mesa, Arizona
  - Horizon Clinical Research Associates, Mesa, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Sagebrush Medical Plaza, Department of Family Medicine, Bakersfield, California
  - Family Medical Center, Foothill Ranch, California
  - Prime-Care Clinical Research, Mission Viejo, California
  - Encompass Clinical Research, Spring Valley, California
  - Orange County Research Center, Tustin, California
  - Quality Care Medical Center, Vista, California
  - Arapahoe Internal Medicine, Littleton, Colorado
  - Institute Diabetes and Metabolic Disease, Newark, Delaware
  - Alliance Medical Reserach Group, Inc., Clearwater, Florida
  - Personal Physician Care, Delray Beach, Florida
  - Century Clinical Research, Inc, Holly Hill, Florida
  - Innovative Research of West Florida, Largo, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Executive Health and Research Associates, Inc., Atlanta, Georgia
  - Capital City Family Medicine, Boise, Idaho
  - Orthopedic Health Care Clinic, Boise, Idaho
  - Sonora Clinical Research, Boise, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Chicago Research Center, Inc., Chicago, Illinois
  - Heart of America Research, Shawnee, Kansas
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Acadia Clinical Research, LLC, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Professional Clinical Reserach -Great Lakes Family Care, Cadillac, Michigan
  - Synergy Medical Education Alliance, Saginaw, Michigan
  - Medex Healthcare Research, Inc, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - Specialty Medical Center, Pahrump, Nevada
  - Bassett Healthcare, Cooperstown, New York
  - DiGiovanna Family Care Center, Great Neck, New York
  - United Physicians Group - Endocrine Division, Great Neck, New York
  - Winthrop University Hospital, Mineola, New York
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Fallen Timbers Internal Medicine LLC, Maumee, Ohio
  - COR Clinical Reserch, LLC, Oklahoma City, Oklahoma
  - Cllinical Research Consultants, Medford, Oregon
  - Covance Clinical Research Unit, Inc, Portland, Oregon
  - Michael A. Azorr, M.D., Portland, Oregon
  - Keystone Clinical Solutions, Altoona, Pennsylvania
  - Southeastern PA Medical Institute, Havertown, Pennsylvania
  - Greenand Seidner Family Practice, Lansdale, Pennsylvania
  - Thomas Jefferson University Div of Endocrinology, Philadelphia, Pennsylvania
  - Founders Medical Practice, Philadelphia, Pennsylvania
  - Research Endeavors, Pittsburgh, Pennsylvania
  - Hillcrest Clinical Research LLC, Simpsonville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - John Joseph, MD PA, Carrollton, Texas
  - Renaissance Clinical Research, Dallas, Texas
  - MCA Research, Houston, Texas
  - Southwest Houston Research, LTD, Houston, Texas
  - Professional for Clinical Research, Plano, Texas
  - Research Across America, Plano, Texas
  - Benjamin Garwood Research, San Antonio, Texas
  - WellMed at Northern Hills, San Antonio, Texas
  - Diabetes and Glandular Disease Research Associates, San Antonio, Texas
  - Diabetes and Glandular Disease - Westside office, San Antonio, Texas
  - Liberty Research Center, Tacoma, Washington
  - Hyperion Clinical Trials, Inc., Charleston, West Virginia